CLINICAL TRIAL: NCT01842828
Title: E-Cigarettes as an Addition to Multi-component Treatment for Tobacco Dependence: A Pilot Study
Brief Title: UK-Czech E-cigarette Study
Acronym: (SUKCES)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: QMUL201208b
Record Dates: First submitted 2013-04-23; First posted 2013-04-30 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2016-02

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Standard of Care; Electronic Nicotine Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care plus electronic cigarettes (Active Comparator): Standard care for smoking cessation plus electronic cigarettes
  Interventions: Other: Standard care plus electronic cigarettes
- Standard care (Other): Standard care for smoking cessation
  Interventions: Other: Standard care plus electronic cigarettes; Behavioral: Standard care

INTERVENTIONS:
Other: Standard care plus electronic cigarettes
Behavioral: Standard care
  Arms: Standard care

SUMMARY:
Currently available smoking cessation treatments help only about 15% of smokers to quit long-term. These treatments do not typically address the behaviours and sensations associated with the act of smoking (e.g. handling a cigarette, inhaling, taste and feel of smoke on the throat). There is evidence that these elements influence smoking behaviour and cessation. Electronic cigarettes (EC) are a new product with a strong potential to be a realistic behavioural replacement for smoking.

Whilst EC deliver nicotine, their use does not involve tobacco combustion, which is the primary source of the many thousands of dangerous chemicals to which smokers of conventional cigarettes are exposed. Studies on EC products and users indicate there is little doubt that they are substantially safer than conventional cigarettes.

The investigators plan to conduct a study one of the very first studies to test the effects of adding EC to standard care on long-term validated outcomes. Before launching such a large and demanding trial however, data are needed on what proportion of smokers would be interested in using EC and what compliance with EC use can be expected, and no data exist to inform how large a sample is needed. This pilot study would provide such data.

A total of 200 smokers would be recruited at smoking cessation clinics in London and Prague. Half the smokers would be randomised to receive standard smoking cessation behavioural support and medication (standard care; SC), and half to receive SC plus EC. The EC group would receive a four week supply of EC. The outcome measures for the study would be smoking status at 4 and 24 weeks after the target quit date, EC use, acceptability, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Smokers who want help with quitting
* Aged 18 or over

Exclusion Criteria:

* Pregnancy, breastfeeding, planning to conceive in the next 6 months
* Enrolled in other research
* Currently using electronic cigarettes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2013-12; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Carbon monoxide (CO)-validated continuous abstinence rates at 4 weeks post-TQD | Four weeks

SECONDARY OUTCOMES:
Carbon monoxide (CO)-validated abstinence rates at 24 weeks post-TQD | Four weeks
Ratings of cigarette withdrawal at 1 and 4 weeks post-TQD | Four weeks
Electronic cigarette use | 24 weeks
Electronic cigarette taste and satisfaction in comparison to conventional cigarettes | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hajek, PhD, Principal Investigator — Queen Mary University of London
Locations (1):
- Tobacco Dependence Research Unit, Queen Mary University of London, London, United Kingdom